CLINICAL TRIAL: NCT01891487
Title: Safety and Efficacy of Bimatoprost 0.03% Solution for the Treatment of Eyebrow Hypotrichosis: A Phase 4 Investigator Initiated Study
Brief Title: Safety and Efficacy of Bimatoprost 0.03% Solution for the Treatment of Thinning Eyebrows
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ATS Clinical Research (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATSBROW-001
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Hypotrichosis
Keywords: Eyebrow; Hypotrichosis; Thinning; Bimatoprost
MeSH Terms: conditions — Hypotrichosis | interventions — Bimatoprost; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Track A (Active Comparator): Those on active study medication
  Interventions: Drug: Track A
- Track B (Placebo Comparator): Those on placebo.
  Interventions: Drug: Track B

INTERVENTIONS:
Drug: Track A — Bimatoprost 0.03% solution applied to eyebrow
  Other Names: Active study drug; Bimatoprost 0.03% solution
  Arms: Track A
Drug: Track B — Refresh Tears applied to eyebrows
  Other Names: Placebo control group; Refresh Tears
  Arms: Track B

SUMMARY:
This is a study researching the safety and efficacy of Bimatoprost 0.03% soultion versus placebo applied to the eyebrow for the treatment of thinning eyebrows. This is a 36 week study where Bimatoprost 0.03% solution/placebo will be applied once daily to the subjects eyebrow for duration of the study.

DETAILED DESCRIPTION:
A parallel, placebo-controlled, single-center, prospective, randomized, double blind, pilot trial to demonstrate bimatoprost 0.03% efficacy in eyebrow hypotrichosis in otherwise healthy individuals with thinning eyebrows. Bimatoprost 0.03% or placebo will be applied to the eyebrow margin once daily for 36 weeks. Adverse events will be assessed, and subjects will complete outcomes questionnaires at study visits. Eyebrow growth and darkening will be scored by the investigator and photography will be taken at each study visit.

Eyebrows are generally composed of three types of hairs: fine vellus hairs are the smallest, with the second type slightly larger, lightly pigmented hairs. The supercilia are the large terminal hairs which are the most visible and are primarily responsible for color and shape of the brow. Eyelashes are composed of terminal hairs, and it has been well demonstrated that bimatoprost application on these hairs will render them longer, thicker and darker (Allergan Protocol 192024-032). It has also been demonstrated that bimatoprost will darken vellus hair, making them more visible. It may be that administering bimatoprost to the eyebrows will cause the terminal hair to become longer, thicker and darker, and make the vellus and lightly pigmented hairs become more noticeable, thus increasing the intensity and fullness of the entire brow.

Multiple studies have been conducted to assess the safety and efficacy of the application of bimatoprost solution to the eyelid for growth of natural eyelashes (Yoelin S, et al, 2010). In 2 active-controlled phase 3 studies for LUMIGAN®, eyelash growth was reported as an adverse event after 3 months of treatment of subjects receiving bimatoprost once daily (Allergan Studies 192024-008 and 192024-009). The application of bimatoprost solution to the eyelid has proven to be effective in enhancing eyelash growth in women when applied daily for 12 weeks (Cohen JL, 2010).

This drug effect has been formally acknowledged in the LUMIGAN® package insert (Appendix 5.2) further supporting the bimatoprost's effect on eyelash growth. The package insert indicates that LUMIGAN® may gradually change eyelashes with regard to increased length, thickness, pigmentation, and number of eyelashes. Since its US approval in 2001, several adverse events of "growth of eyelashes" have been reported in conjunction with the use of LUMIGAN®.

Subjects will be randomized to Track A, active study drug, bimatoprost 0.03% solution, or to Track B, placebo. Each track will apply the same dose, 1 drop per eyebrow once daily, to determine the safety and efficacy of bimatoprost 0.03% solution versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Females and males, ages 18-75 years with brows that are naturally thinning with a score of 1 (very thin) or 2 (thin) at baseline as determined by the Investigator Global Eyebrow Assessment (IGEA).
* Subjects who agree to forgo any additional treatment to the brows, such as waxing, plucking, threading and/or tinting for the duration of the study.
* Desires to participate in a research study

Exclusion Criteria:

* Any uncontrolled systemic disease.
* Any known diseases or abnormalities to the eyelid or eyebrow.
* Known allergies or reactions to bimatoprost or placebo ingredients.
* Pregnancy.
* Subjects that have thinning brows as a result of over plucking, trichotillomania, chemotherapy or any other condition or treatment that causes hair loss.
* Subjects who have used any over the counter or prescription eyebrow growth product 3 months prior to baseline.
* Subjects with tattooed eyebrows and/or any permanent or semi-permanent tint or dye within 3 months prior to baseline.
* Subjects with a score of 3 or 4 on the eyebrow scale.
* Current enrollment in an investigational drug or device study or participation in such a study 30 days prior to baseline.
* Subjects using prostaglandin analogs for the treatment of high intraocular pressure.
* Aphakic subjects and/or pseudophakic subjects with a torn posterior lens capsule.
* Subjects with known risk factors for macular edema.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
One grade improvement at week 16, 24 and 36 as based on the IGEA | Week 16, 24 and 36
  Target area of both left and right eyebrow will be examined for a one grade improvement based on the Investigator Global Eyebrow Assessment (IGEA) (section 17 of protocol) at baseline, week 16, 24 and 36 for Track A and Track B subjects. Target area is delineated by the mid-pupillary line to the lateral canthus.

SECONDARY OUTCOMES:
Grade improvement based on IEA4 at week 16, 24 and 36 | Week 16, 24 and 36
  Intensity (defined as thickness, darkness and hair quantity) of the target area of both left and right eyebrow based on the Investigator Eyebrow Assessment 4 Point Brow Scale at baseline, week 16, 24 and 36 for Track A and Track B subjects. Subject satisfaction with their brows (PRO measure) at week 36 for Track A Track B. Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ava Shamban, MD, Principal Investigator — ATS
Locations (1):
- Ava MD, Santa Monica, California, United States

REFERENCES:
- [Background] Allergan Protocol 192024-032, June 2008 Safety and Efficacy of Bimatoprost Solution in Increasing Overall Eyelash Prominence.
- [Result] Allergan Protocol 192024-008 A multicenter, double-masked, randomized, parallel, three-month study (with treatment extended to one year) of the safety and efficacy of ANG 192024 0.03% ophthalmic solution, administered once- daily or twice-daily compared with timolol 0.5% ophthalmic solution administered twice-daily, in subjects with glaucoma or ocular hypertension [12 month report].
- [Result] Allergan Protocol 192024-009 A multicenter, double-masked, randomized, parallel, three-month study (with treatment extended to one year) of the safety and efficacy of ANG 192024 0.03% ophthalmic solution administered once-daily or twice daily compare with timolol 0.5% ophthalmic solution administered twice-daily, in subjects with glaucoma or ocular hypertension [12 month report].
- [Result] Cohen JL. Enhancing the growth of natural eyelashes: the mechanism of bimatoprost-induced eyelash growth. Dermatol Surg. 2010 Sep;36(9):1361-71. doi: 10.1111/j.1524-4725.2010.01522.x. PMID 20384750
- [Result] Yoelin S, Walt JG, Earl M. Safety, effectiveness, and subjective experience with topical bimatoprost 0.03% for eyelash growth. Dermatol Surg. 2010 May;36(5):638-49. doi: 10.1111/j.1524-4725.2010.01519.x. Epub 2010 Apr 1. PMID 20384751